CLINICAL TRIAL: NCT03178435
Title: Preventing Acute Kidney Injury and Improving Outcome in Critically Ill Patients Utilising Risk Prediction Score - a Pilot Feasibility Randomized Controlled Trial
Brief Title: Preventing Acute Kidney Injury and Improving Outcome in Critically Ill Patients Utilising Risk Prediction Score
Acronym: PRAIOC-RISKS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Tarek Samy Abdelaziz, Senior lecturer, Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: KA-13050
Record Dates: First submitted 2017-06-04; First posted 2017-06-07 (Actual); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Acute Kidney Injury; Critical Illness
Keywords: risk score; Acute kidney injury; critical care
MeSH Terms: conditions — Acute Kidney Injury; Critical Illness

STUDY DESIGN:
Intervention Model Description: interventional cluster randomised trial -pilot /feasibility study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Observational (No Intervention): patients will be recruited to this arm to observe prospectively the incidence of AKI among critically ill patients.patients will receive the standard care.No other intervention will be delivered
- Interventional (Active Comparator): Patients in this arm will be subject to AKI risk score. This risk score was recently developed and validated in Mayo clinic the intervention will be Measures to prevent AKI among critically ill patients
  Interventions: Other: Measures to prevent AKI among critically ill patients

INTERVENTIONS:
Other: Measures to prevent AKI among critically ill patients — 1. Meticulous optimization of the fluid balance
  2. Avoidance of nephrotoxic medications where possible
  3. Optimisation of the hemodynamic status
  4. Avoidance of blood transfusion unless marked acute blood loss or symptomatic anemia
  5. Optimization of the underlying medical condition
  6. Seek expert renal advise when necessary
  Arms: Interventional

SUMMARY:
An interventional controlled trial to test the feasibility of applying risk score based prevention for critically ill patient at high risk to develop acute kidney injury (AKI)

DETAILED DESCRIPTION:
Background and rationale AKI is common in the intensive care unit .It contributes significantly to mortality and morbidity .the estimated incidence or AKI among critically ill patients is 30-40% and morality is high.

There is a well recognized gap between the optimal care and the delivered care regarding prevention and management of AKI.

The focus over the last few years has been on early detection. A panel of urinary biomarkers have proved helpful for early detection of AKI. However the cost and low specificity make no single one of them solely reliable .using a panel of bio-markers increases their specificity.

The concept of electronic alerts has been recently introduced. Some trials have been testing its impact on the outcome of AKI. The benefit of electronic alerts is still uncertain .A meta-analysis is currently underway to synthesize stronger evidence of electronic alerts benefit.

Another evolving area, is the development of risk score to predict AKI and and hence applying timely preventive measures.

KDIGO recommends applying preventive measures to high risk patients. However no study to date has tested risk scores based interventions

Hypothesis:

We will use the recently validated score to predict AKI in ICU patients. We will then apply preventive measures. To patients at risk .To our knowledge this is the first study to apply preventive interventions based on AKI risk score assessment

ELIGIBILITY:
Inclusion Criteria:

All adult patients (≥18 year old) admitted to the intensive care unit and do not fulfill the criteria for the diagnosis of AKI by Kidney Disease Improving Global Outcome (KDIGO) definition

Exclusion Criteria:

1. Patients who have already developed AKI at the time of intensive care unit ICU admission.
2. Patients with insufficient medical records to obtain previous medical history
3. Patients who lack mental capacity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-04-01 (Actual); Study Completion 2018-09-01 (Actual)

PRIMARY OUTCOMES:
Incidence of AKI | during 7 days of ICU admission
  We will compare the incidence rate between the interventional and the observational arm

SECONDARY OUTCOMES:
30 day mortality | 30 days
  all cause mortality during 30 days of ICU admission or within 30 days of developement of AKI
Time to recovery after development of AKI | 30 days
  Time interval between the diagnosis of AKI and recovery of either blood chemistry or oliguria
Deterioration of AKI stage | 30 days
  Transition from initial stage KDIGO stage 1 to either 2 or 3 .Transition from initial stage 2 to 3
Duration of dialysis dependency | 30 days
  time patient remains dialysis-dependant after severe AKI.

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo university hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No